CLINICAL TRIAL: NCT00464464
Title: Treating Depression in Parkinson's Disease: A New Method
Brief Title: Coping With Depression in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0220060139
Record Dates: First submitted 2007-04-20; First posted 2007-04-23 (Estimated); Results first posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Parkinson's Disease; Depression
Keywords: Parkinson's disease; PD; depression; cognitive-behavioral therapy; social support
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): cognitive-behavioral therapy
  Interventions: Behavioral: cognitive-behavioral therapy
- 2 (No Intervention): standard medical care

INTERVENTIONS:
Behavioral: cognitive-behavioral therapy — The therapy will consist of 10 weekly individual cognitive-behavioral treatment sessions, lasting 1 hour each and modified to meet the unique needs of each individual with PD.
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the efficacy of a cognitive-behavioral treatment, that includes a caregiver-focused social support intervention, for depression in persons with Parkinson's disease.

Individuals who are unable to travel to the study site, but are interested in participating and meet all other eligibility requirements, will be allowed to participate over the phone.

DETAILED DESCRIPTION:
Depression is the most common emotional problem found in persons with Parkinson's disease (PD). It causes immense personal suffering and is associated with increased disability and burden to caregivers. Despite the adverse consequences of depression in PD, there are virtually no studies to guide clinical treatment. Several studies are currently examining the effectiveness of antidepressant medication for depression in PD. However, there have been no studies to examine the effectiveness of non-medication approaches, such as cognitive-behavioral therapy, despite the success of these techniques in other populations. Cognitive-behavioral therapy teaches people with PD to become more aware of their thoughts and feelings and to change thinking patterns and behaviors that may be related to symptoms of depression.

The purpose of this study is to determine if cognitive-behavioral therapy--with a caregiver-focused social support intervention--is effective in treating depression in persons with PD. This study will enroll 80 people with PD and their caregivers. Forty participants with PD will be randomly chosen to receive the study treatment in addition to standard medical care. The other 40 will only receive standard medical care and will have the option to receive the study treatment after completing all study assessments (4 months after the initial evaluation).

The study treatment will consist of 10 weekly individual cognitive-behavioral treatment sessions, lasting 1 hour each and modified to meet the unique needs of each individual with PD. Caregivers will attend 4 separate educational sessions-lasting 30 minutes each--designed to provide them with the tools needed to reinforce and supplement the material presented in the cognitive-behavioral sessions. Duration of the study for participants is 15 weeks.

This is the first study to evaluate the impact of a cognitive-behavioral treatment for PD depression in a randomized controlled trial. Information gained from this study may be beneficial in treating depression in persons with PD.

ELIGIBILITY:
Persons with PD Inclusion Criteria:

* Confirmed diagnosis of PD with no significant motor fluctuations or dementia.
* Major Depression, Dysthymia, or Depression NOS (Clinically significant depression not otherwise specified).
* 35-85 years old.
* Willingness to ask a family member or friend, with whom the patient has regular contact, to be involved in treatment.
* Patients will be allowed to remain on antidepressant medications that have been stabilized (e.g., no dose changes) for at least 6 weeks prior to screening provided that they do not have plans to change these medications while in the study.
* Patients will be allowed to remain on sedative-hypnotics or anxiolytics that have been stabilized for at least 4 weeks prior to screening. Patients who are taking these medications at screening and qualify for participation will be asked to remain on a stable course of these medications throughout the trial.
* Taking a stable dose of dopaminergic replacement therapy for at least one month

Persons with PD Exclusion Criteria:

* DSM-IV criteria for a psychotic disorder, bipolar disorder, organic brain syndrome, or psychoactive substance dependence or abuse (Nicotine or caffeine dependence is allowed). Other psychiatric co-morbidity is not exclusionary as long as the depressive disorder is primary.
* Active suicidal ideation.
* An unstable major medical condition that would interfere with the study.
* Plans to engage in additional psychotherapy during the study (PD support group is ok).
* A diagnosis of dementia, defined as above.
* Significant motor fluctuations, defined as above; mild end of dose wearing off is allowed.
* Patients unwilling or unable to maintain a stable dose of dopaminergic replacement therapy during the trial.
* Use of mood-stabilizers or antipsychotic medication.

Caregiver Inclusion Criteria:

* Ages 25 to 85
* Daily contact with a friend, family member, or spouse with depression and PD *MMSE > 26 [Mini Mental Status Exam score of greater than 26 (i.e., no signs of significant memory impairment)].

Caregiver Exclusion Criteria:

* Active suicidal ideation
* An unstable major medical or psychiatric condition
* Evidence upon clinical interview of substance abuse/dependence

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roseanne D Dobkin, PhD, Principal Investigator — Associate Professor of Psychiatry Rutgers-Robert Wood Johnson Medical School; Matthew Menza, MD, Study Chair — Professor and Chair, Department of Psychiatry, Rutgers- Robert Wood Johnson Medical School (Primary Mentor)
Locations (1):
- Rutgers, Robert Wood Johnson Medical School, 675 Hoes Lane, Room D-317, Piscataway, New Jersey, United States

REFERENCES:
- [Result] Dobkin RD, Menza M, Allen LA, Gara MA, Mark MH, Tiu J, Bienfait KL, Friedman J. Cognitive-behavioral therapy for depression in Parkinson's disease: a randomized, controlled trial. Am J Psychiatry. 2011 Oct;168(10):1066-74. doi: 10.1176/appi.ajp.2011.10111669. Epub 2011 Jun 15. PMID 21676990
- [Result] Dobkin RD, Rubino JT, Allen LA, Friedman J, Gara MA, Mark MH, Menza M. Predictors of treatment response to cognitive-behavioral therapy for depression in Parkinson's disease. J Consult Clin Psychol. 2012 Aug;80(4):694-9. doi: 10.1037/a0027695. Epub 2012 Mar 12. PMID 22409644
- [Result] Dobkin RD, Menza M, Allen LA, Tiu J, Friedman J, Bienfait KL, Gara MA, Mark MH. Telephone-based cognitive-behavioral therapy for depression in Parkinson disease. J Geriatr Psychiatry Neurol. 2011 Dec;24(4):206-14. doi: 10.1177/0891988711422529. PMID 22228827
- [Result] Dobkin RD, Troster AI, Rubino JT, Allen LA, Gara MA, Mark MH, Menza M. Neuropsychological outcomes after psychosocial intervention for depression in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 2014 Winter;26(1):57-63. doi: 10.1176/appi.neuropsych.12120381. PMID 24275895
- [Result] Dobkin RD. The relationship between telephone-administered cognitive-behavioral therapy for depression and neuropsychological functioning in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 2014 Apr 1;26(2):E10-1. doi: 10.1176/appi.neuropsych.13030065. PMID 24763770
- [Derived] Dobkin RD, Mann SL, Interian A, Gara MA, Menza M. Cognitive behavioral therapy improves diverse profiles of depressive symptoms in Parkinson's disease. Int J Geriatr Psychiatry. 2019 May;34(5):722-729. doi: 10.1002/gps.5077. Epub 2019 Mar 4. PMID 30714202

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive-Behavioral Therapy Condition: Participants in the "Cognitive-Behavioral Therapy" condition will receive 10 weekly individual cognitive-behavioral treatment sessions, lasting one hour each and modified to meet the unique needs of each individual with PD.
  These participants will also receive clinical monitoring of their depressive symptoms at 4 points during the trial and once a month after the trial has ended. During the trial, these participants will continue medical or psychiatric care they had been receiving regularly for 6 or more weeks prior to entering the trial.
- Standard Medical Care Condition: Participants in the "Standard Medical Care" condition will receive clinical monitoring of their depressive symptoms at 4 points during the trial and once a month after the trial ended. These participants will continue medical or psychiatric care they had been receiving regularly for 6 or more weeks prior to entering the trial, but will not be given any new therapy during the trial.
Period: Overall Study
Arm/Group | Cognitive-Behavioral Therapy Condition | Standard Medical Care Condition
Started | 41 | 39
Completed | 36 | 36
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive-Behavioral Therapy Condition | Standard Medical Care Condition | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.73 (9.89) | 65.44 (11.23) | 64.56 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 38 | 36 | 74
  African American | 0 | 1 | 1
  Asian | 3 | 1 | 4
  Pacific Islander | 0 | 1 | 1
  Hispanic | 2 | 1 | 3
  Non-Hispanic | 39 | 38 | 77
Parkinson's disease duration [Mean (Standard Deviation); unit: years] | 6.53 (5.53) | 6.13 (5.56) | 6.34 (5.51)
Dementia Rating Scale score [Mean (Standard Deviation); unit: units on a scale] — The Dementia Rating Scale - 2 (DRS-2) was used to assess severity of symptoms associated with dementia in study participants. The measure includes sub-scales addressing Attention (ATT), Initiation/Perseveration (I/P), Construction (CONST), Conceptualization (CONCEPT), and Memory (MEM).
  The total score (a sum of the five sub-scale scores) was used as the outcome measure value. Possible DRS total scores range from 0 to 144, with higher values representing more severe dementia symptomatology, and lower scores representing less severe dementia symptomatology.
  units on a scale | 139.44 (3.8) | 136.97 (5.5) | 138.24 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale: Baseline
Description: This measure uses the Hamilton Depression Rating Scale (HDRS) to express the average severity of depressive symptoms for a) all participants in the Cognitive-Behavioral Therapy condition and b) all participants in the Standard Medical Care condition, at the outset of the trial.
  The total score on the HDRS (range = 0 to 84) was used as the outcome measures value, with higher values indicating more severe depressive symptomatology and lower scores representing less severe depressive symptomatology.
Time Frame: 0 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioral Therapy Condition | Standard Medical Care Condition
Number analyzed (Participants) | 41 | 39
units on a scale | 20.93 (4.56) | 19.38 (4.56)

2. Primary Outcome: Hamilton Depression Rating Scale: Midpoint
Description: This measure uses the Hamilton Depression Rating Scale (HDRS) to express the average severity of depressive symptoms for a) all participants in the Cognitive-Behavioral Therapy condition and b) all participants in the Standard Medical Care condition, after 5 weeks of the trial.
  The total score on the HDRS (range = 0 to 84) was used as the outcome measures value, with higher values indicating more severe depressive symptomatology and lower scores representing less severe depressive symptomatology.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioral Therapy Condition | Standard Medical Care Condition
Number analyzed (Participants) | 41 | 39
units on a scale | 14.92 (4.73) | 19.71 (4.56)

3. Primary Outcome: Hamilton Depression Rating Scale: Endpoint
Description: This measure uses the Hamilton Depression Rating Scale (HDRS) to express the average severity of depressive symptoms for a) all participants in the Cognitive-Behavioral Therapy condition and b) all participants in the Standard Medical Care condition, at the end of the 10 week trial.
  The total score on the HDRS (range = 0 to 84) was used as the outcome measures value, with higher values indicating more severe depressive symptomatology and lower scores representing less severe depressive symptomatology.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioral Therapy Condition | Standard Medical Care Condition
Number analyzed (Participants) | 41 | 39
units on a scale | 13.58 (4.72) | 19.33 (4.55)

4. Primary Outcome: Hamilton Depression Rating Scale: Follow-Up Evaluation
Description: This measure uses the Hamilton Depression Rating Scale (HDRS) to express the average severity of depressive symptoms for a) all participants in the Cognitive-Behavioral Therapy condition and b) all participants in the Standard Medical Care condition, 4 weeks after the trial ended.
  The total score on the HDRS (range = 0 to 84) was used as the outcome measures value, with higher values indicating more severe depressive symptomatology and lower scores representing less severe depressive symptomatology.
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive-Behavioral Therapy Condition | Standard Medical Care Condition
Number analyzed (Participants) | 41 | 39
units on a scale | 14.52 (4.75) | 19.31 (4.63)

ADVERSE EVENTS:
Arm/Group | Cognitive-Behavioral Therapy Condition | Standard Medical Care Condition
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes